CLINICAL TRIAL: NCT06837298
Title: The Effect of Vicia Faba Hydrolysate Supplementation on Muscle Strength Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2414
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Muscle Damage; Muscle
Keywords: DOMS; exercise; damaging; muscle; muscle recovery; vicia faba; fava bean; PeptiStrong
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): PeptiStrong® capsules 2.4 grams per day for 17 days
  Interventions: Other: Placebo control capsules
- PeptiStrong® 17 days (Experimental): PeptiStrong® capsules 2.4 grams/day for 17 days
  Interventions: Other: PeptiStrong® supplement capsules with same appearance as placebo capsules
- PeptiStrong® 3 days (Experimental): 14 days of Placebo followed by 3 days of PeptiStrong®
  Interventions: Other: PeptiStrong® supplement capsules following muscle damaging exercise on Day 14

INTERVENTIONS:
Other: Placebo control capsules — 2.4 grams (g) daily
  Arms: Placebo
Other: PeptiStrong® supplement capsules with same appearance as placebo capsules — 2.4 g daily
  Arms: PeptiStrong® 17 days
Other: PeptiStrong® supplement capsules following muscle damaging exercise on Day 14 — 2.4 g placebo capsules for 14 days, then 3 days 2.4 g of PeptiStrong® capsules following one muscle damaging exercise session
  Arms: PeptiStrong® 3 days

SUMMARY:
To investigate the effect of Vicia faba protein concentrate, a protein derived from Fava bean extract, on delayed onset muscle soreness (DOMS). Participants receive either 2.4g/day of PeptiStrong® supplement capsules or placebo capsules for 14 days until a strenuous exercise session. For the last 3 days, 2/3 of them stay on the same treatment and 1/3 of them switch from placebo to PeptiStrong®.

DETAILED DESCRIPTION:
Delayed onset muscle soreness (DOMS) is the result of eccentric muscle contraction and is caused by small tears in the myofibrils. Damage to the muscle fibers causes pain, inflammation, and reduced range of motion which can delay recovery. Peak effects are often experienced 48 - 72 hours following the exercise session but can last up to 7 days post-exercise. Various modalities are utilized to reduce DOMS such as cryotherapy, massage, and compression. However, nutritional supplements have also been studied including Omega 3 fatty acids, creatine monohydrate, tart cherry juice, vitamin D, and probiotics.

A recent study (Kerr, et al., 2023) investigated the effects of a protein supplement (PeptiStrong®) from Vicia faba protein concentrate, a protein derived from Fava bean extract. Results showed that 17 days of 2.4 grams of PeptiStrong® significantly improved muscle strength, reduced muscle fatigue, and reduced myostatin expression during the 72 hour recovery period compared to placebo following a strenuous bout of eccentric exercise. This study aims to repeat the methods of Kerr, et al. with the addition of females and a third experimental group. In addition to 17 days of supplementation with Vicia faba Hydrolysate or placebo, a third group will be given 14 days of placebo followed by 3 days of the Vicia faba Hydrolysate supplement to determine if short-term supplementation results in a similar benefit.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 45 years of age.
* Willing to fast overnight on the 4 testing occasions.
* Participants agree to abstain from taking additional supplements throughout the testing period, with particular emphasis placed upon protein-based products (e.g., whey or casein based protein powders; animal derived protein hydrolysates; natural supplements constituted of vegetative protein hydrolysates from rice, fava bean, pea, carrot, spirulina, broccoli, potatoes; marine derived secondary metabolite products or protein hydrolysates including Omega-3 capsules or DHA).
* Moderately active (exercise 3-5 days per week)
* Fluent in reading, writing, and speaking English
* Participants agree to maintain their normal diet and perform only light to moderate exercise for the duration of the study.
* BMI between 18.5 and 29.9 kg/m2
* Participants agree to refrain from consuming alcohol in the 48 hours leading up to a test day.
* Willingness to complete questionnaires, records and diaries associated with the study and to complete all lab visits.
* Refrain from any exercise from 48 hours prior to each test or blood draw.
* Healthy as determined by General Health Questionnaire.
* Non-smoker

Exclusion Criteria:

* Individuals that are glucose-6-phosphate-dehydrogenase deficient. The test product in this study contains fava bean extract which may produce favism in genetically susceptible individuals.
* Alcohol or drug abuse in the past year.3. Testosterone or estrogen supplementation (not including women on oral contraceptives)
* Pregnant or nursing or planning to become pregnant.
* Participation in any other clinical trial in the past 30 days. Participation in any PepsiCo trial in the past 6 months
* Volunteers with unstable medical conditions.
* Any complaints that could interfere with the ability to exercise.
* Individuals who are cognitively impaired or unable to give informed consent.
* Any co-morbidities interacting with mobility or muscle metabolism of the lower limbs (e.g. arthritis, spasticity / rigidity, all neurological disorders, paralysis).
* Creatine supplements, corticosteroids, NSAIDS, amino acids, injectible peptides, collagen, and nicotinamide (Vit B3/niacin).
* Presence or history of neurological disorders or significant psychiatric illness.
* Any condition the study investigator believes would interfere with eligibility following the study protocol, effect the study results, or put the subject at undue risk.
* Participation in resistance or aerobic exercise within 48 hours of the test days.
* Participation of >3 high-intensity exercise sessions per week.
* Undertake recovery methods such as sea swims, foam rolling, cryotherapy or excessive stretching during days 14-17.
* Have been in contact with a suspected or confirmed case of COVID-19 in previous 14 days.
* Are Hepatitis A- or B-positive or have had a sexual partner infected with hepatitis or HIV and not taking medication.
* Are not employed by, or have a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If you are unsure if a company would be considered a competitor to Gatorade, let the study investigator know the name of the other company and the nature of your relationship to that company before ou sign the informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Concentric knee extension and flexion strength | Following strenuous muscle damaging exercise on Day 14
  Assessed at an angular velocity of 60°/s through the range of 0-100° knee flexion using an isokinetic dynamometer (Biodex)

SECONDARY OUTCOMES:
Exercise induced expression of markers of muscle stress | Days 14 at Baseline and 2 hrs post strenuous exercise, and on Days 16 and 17 at 10 minutes post exercise
  Plasma concentrations of IL-6, IL-15, fractalkine, irisin, FGF21, myostatin, osteocrin / PEP- 2414 Page 9 of 32 1/29/25 V6 musclin, osteonectin/SPARC
Ratings of soreness, fatigue, pain, and tenderness. | Days 14, 15, 16, 17 based on the previous 24 hours
  Rated on a 4-item Recovery survey, anchored from none to extreme
Fatigue index | Baseline Day 0, Day 16 and Day 17 for each strength test
  Calculated from the strength tests using the following equation: (highest force - lowest force) / highest force

CONTACTS AND LOCATIONS:
Overall Officials: Kris Osterberg, PhD, RD, Principal Investigator — PepsiCo R&D Life Sciences, Sports Science
Locations (1):
- Gatorade Sports Science Institute at IMG Academy, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No